CLINICAL TRIAL: NCT03784456
Title: Impact of Increased Protein Density Diet to Muscle Mass and Strength Among Mid-aged and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Laurel Corporation, Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-001-A-2
Record Dates: First submitted 2018-12-06; First posted 2018-12-24 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Muscle Loss; Muscle Weakness; Fragility
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: This program is designed as a double blind parallel randomized intervention. The primary purpose of this program is Prevention.
Who Masked: Participant
Masking Description: The program is designed as a double blind test, randomized intervention. Which meant that neither the subjects nor the PI and co-PI would not know which kind of diet they're going to obtain. Only investigators and test provider would know the meals corresponding to respective groups of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25% protein group (Experimental): This experimental arm will be given meals containing 25% protein under same estimated calorie menus and protein may come from either egg, meat, fish, soy, or milk product. The meals would be provided 2 times per day, 5 days per week. The program will last for 12 weeks.
  Interventions: Dietary Supplement: 25% protein
- 15% protein group (Active Comparator): This control arm will be given meals containing 15% protein under same estimated calorie menus and protein may come from either egg, meat, fish, soy, or milk product. The meals would be provided 2 times per day, 5 days per week. The program will last for 12 weeks.
  Interventions: Dietary Supplement: 15% protein

INTERVENTIONS:
Dietary Supplement: 25% protein — Compared to usual group of 15% protein in meals, intervention group will receive 25% protein contents under same estimated calorie menus. Protein may come from either egg, meat, fish, soy, or milk product.
  Arms: 25% protein group
Dietary Supplement: 15% protein — Designed as comparator , compared to empirical arm of 25% protein in meals, intervention group will receive 15% protein contents under same estimated calorie menus. Protein may come from either egg, meat, fish, soy, or milk product.
  Arms: 15% protein group

SUMMARY:
The subjects of this intervention program are mainly based on community-dwelling mid-aged and older adults. The investigator's program will provide meals containing different proportionated protein.As this project is a double blind test, only the investigators will know which subject corresponding to specific group of diets.

Besides, the investigators use the valued-based healthcare standard set as well as the Center for Epidemiological Studies-Depression, Charlson's comorbidity index Montreal Cognitive Assesment ,and Mini Nutritional Assessment as outcome measures and to use the randomized controlled trial design to validate if increased protein density diet could improve the vitality and health of mid-aged and old adults .

DETAILED DESCRIPTION:
With aging, functions of every organs become to decline. Muscle mass, is one of the decline. According to previous research, adults would lose 40% among from aged 20 to 70. If muscle mass decline combining with the decline of muscle strength is so called Sarcopenia.When muscle mass decline, infectious risk gets higher, and resilience after illness gets lower. In addition, activity and life quality are also responsible for falling, cognitive difficulty, disability and mortality among seniors. We hope to find out the etiologies of Sarcopenia through this program and develop prevention strategy and model to mollify the the negative effect of rapid aging society.

ELIGIBILITY:
Inclusion Criteria:

* People who aged 40-75 years
* Patients with following characteristics:
* feeling loss in activity
* detecting decline in self's walking speed.
* feeling tired of doing everything.
* having fell in last year.
* People can accept undergoing MRI
* People willing to follow the program and cooperate with us for following tracking.
* People who are neither vegan nor vegetarian
* People agree and be able to sign the informed consent.

Exclusion Criteria:

* People cannot intake provided meals (e.g.: vegans or vegetarians) or any other who is allergic to our diets.
* People with any disease affecting their limbs, including:
* having fracture on limbs in the past 6 months
* having severe arthritis in the past 6 months
* any other whom PI recognized as weak control of their nervous system( e.g.: Parkinson's disease and stroke).
* People with intermittent limp caused by peripheral artery diseases
* People with weak control of mental disorder
* People with weak control of Cardiopulmonary disease
* People with weak control of Malignant tumor
* People with weak control of kidney diseases (eGFR <60ml/min/1.73)
* People with Visual impairment and Hearing disorder which cannot help to complete the program.
* People who are unable to undertake MRI
* People who have underwent hormone treatment and planned to undergo hormone treatment during program session.
* Any other condition that PI recognized as not suitable

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline muscle strength after 12 weeks | baseline,12 weeks
  measured by hand grip
Changes form baseline QUALITY OF LIFE after 12 weeks | baseline, 12 weeks
  measured by the 36-Item Short Form Health Survey (SF-36), ranged 0-100, higher values represent a better condition
Change from baseline Nutrition intake after 12 weeks | baseline, 12 weeks.
  measured by Mini-nutritional assessment questionnaire. ranged 0-30, higher values represent a better condition
Change from baseline depression after 12 weeks | baseline,12 weeks
  measured by the Center for Epidemiological Studies-Depression (CES-D) ranged 0-60, higher values represent a worse condition
Change from baseline cognitive ability after 12 weeks | baseline, 12 weeks
  measured by Montreal Cognitive Assessment (MoCA) , ranged 0-30, higher values represent a better condition
Change from baseline endurance after 12 weeks | baseline, 12 weeks
  measured by 6-minute walk distance
Change from baseline walking speed after 12 weeks | baseline, 12 weeks
  measured by six-meter walking speed
Change from baseline timed up and go test after 12 weeks | baseline, 12 weeks
  measured by timed up and go test (TUG) and six-meter walking speed

SECONDARY OUTCOMES:
Change from baseline numbers of Complete blood count after 12 weeks | baseline,12 weeks
  Change from baseline numbers of Complete blood count after 12 weeks
Change from baseline concentration of Albumin after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Albumin after 12 weeks
Change from baseline concentration of Alanine Aminotransferase (ALT) after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Alanine Aminotransferase (ALT) after 12 weeks
Change from baseline concentration of Aspartate Aminotransferase (AST) after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Aspartate Aminotransferase (AST) after 12 weeks
Change from baseline concentration of blood urea nitrogen after 12 weeks | baseline,12 weeks
  Change from baseline concentration of blood urea nitrogen after 12 weeks
Change from baseline concentration of Creatinin after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Creatinin after 12 weeks
Change from baseline concentration of Fasting glucose after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Fasting glucose after 12 weeks
Change from baseline concentration of Fasting insulin after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Fasting insulin after 12 weeks
Change from baseline concentration of Total Cholesterol after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Total Cholesterol after 12 weeks
Change from baseline concentration of Triglyceride after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Triglyceride after 12 weeks
Change from baseline concentration of high-density lipoprotein cholesterol after 12 weeks | baseline,12 weeks
  Change from baseline concentration of high-density lipoprotein cholesterol after 12 weeks
Change from baseline concentration of low-density lipoprotein cholesterol after 12 weeks | baseline,12 weeks
  Change from baseline concentration of low-density lipoprotein cholesterol after 12 weeks
Change from baseline concentration of high-sensitivity C-reactive protein after 12 weeks | baseline,12 weeks
  Change from baseline concentration of high-sensitivity C-reactive protein after 12 weeks
Change from baseline concentration of dehydroepiandrosterone after 12 weeks | baseline,12 weeks
  Change from baseline concentration of dehydroepiandrosterone after 12 weeks
Change from baseline concentration of 25-(OH)-Vit. D after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of 25-(OH)-Vit. D after 12 weeks
Change from baseline concentration of Leptin after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of Leptin after 12 weeks
Change from baseline concentration of urine protein after 12 weeks | baseline, 12 weeks
  Change from baseline concentration of urine routine after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, MD.PhD., Principal Investigator — Aging and Health Research Center, National Yang Ming University
Locations (1):
- National Yang Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided